CLINICAL TRIAL: NCT04124809
Title: Truth or Dare; Artificial Blastocoel Collapse of Human Blastocysts Before Vitrification
Brief Title: Truth or Dare; Artificial Blastocoel Collapse Using Laser Before Blastocyst's Vitrification Versus Non-laser Usage
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no fund for recruitment
Sponsor: Benha University (Other)
Collaborators: Hawaa Fertility Center (Other)
Responsible Party: Principal Investigator, Ahmed Saad, Assistant professor of Obstetrics & Gynecology, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Hawaa-7
Record Dates: First submitted 2019-10-08; First posted 2019-10-11 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Blastocyst Disintegration
Keywords: blastocyst; Vitrification; artificial collapse; survival rate
MeSH Terms: conditions — Embryo Loss

STUDY DESIGN:
Intervention Model Description: patients with sibling blastocysts divided into 2 groups: Study group (artificially laser-collapsed blastocysts; n=71) & control group (blastocysts were vitrified without laser collapse; n=66) then reexpansion speed and survival rate was assessed immediately & at 140 min after thawing and compared between two groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: only the investigator knew the procedure provided for each case
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (artificially laser-collapsed blastocysts) (Experimental): laser was used as an intervention before blastocyst vitrification to assist rapid blastocyst collapse with vitrification
  Interventions: Device: laser assisted collapse
- & control group (blastocysts were vitrified, no laser collapse (No Intervention): blastocyst were vitrified without laser assisted collapse

INTERVENTIONS:
Device: laser assisted collapse — Apply 1-2 pulses of laser using the Saturn between 2 adjacent trophectoderm cells away from the inner cell mass in the blastocysts
  Arms: Study group (artificially laser-collapsed blastocysts)

SUMMARY:
: This prospective randomized observational study aimed to compare behavior of artificially collapsed blastocysts to blastocysts that were vitrified without artificial collapse.

DETAILED DESCRIPTION:
One arm study of 60 patients with sibling blastocysts divided into 2 groups: Study group (artificially laser-collapsed blastocysts; n=71) & control group (blastocysts were vitrified without laser collapse; n=66) then reexpansion speed and survival rate was assessed immediately & at 140 min after thawing and compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age limit 20-37 At least 6 good quality blastocysts per case. expansion rate 3-4

Exclusion Criteria:

* bad quality blastocysts expansion rate less than 3

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — blastocysts of infertile couples
Enrollment: 10 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
survival rate | immediately after thawing
  survival rate will be assessed immediately after thawing and compared between both groups.
survival rate | 140 min after thawing
  survival rate will be assessed at 140 minutes after thawing and compared between both groups.

CONTACTS AND LOCATIONS:
Overall Officials: sahar A Eissa, Ph. D, Principal Investigator — HFC
Locations (1):
- Hawaa Fertility Center, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the main individual characters of the blastocysts and he data after warming
Supporting Information: Study Protocol
Time Frame: After publication of the study , for 6 months
Access Criteria: saharafify @yahoo.com